CLINICAL TRIAL: NCT03703882
Title: A Randomized, Double-Blind, Placebo-Controlled, Global Phase 3 Study of Edasalonexent in Pediatric Patients With Duchenne Muscular Dystrophy
Brief Title: Phase III Study of Edasalonexent in Boys With Duchenne Muscular Dystrophy
Acronym: PolarisDMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catabasis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAT-1004-301
Record Dates: First submitted 2018-10-08; First posted 2018-10-12 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Muscular Dystrophies; Musculoskeletal Diseases; Neuromuscular Diseases; Duchenne muscular dystrophy; DMD; dystrophin; dystrophy; Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Musculoskeletal Diseases; Neuromuscular Diseases | interventions — edasalonexent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose 1 (Experimental): Edasalonexent 100 mg/kg/day. Capsules taken by mouth three times per day.
  Interventions: Drug: Edasalonexent
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Edasalonexent — 100 mg/kg/day
  Other Names: Edasa; CAT-1004
  Arms: Dose 1
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The PolarisDMD study is a Phase 3, global study to evaluate the efficacy and safety of edasalonexent in pediatric patients with a genetically confirmed diagnosis of DMD. Male patients from 4-7 years of age (up to 8th birthday) will be enrolled.

Edasalonexent is an orally administered small molecule that inhibits NF-kB, which is the key link between loss of dystrophin and disease pathology and plays a fundamental role in the initiation and progression of skeletal and cardiac muscle disease in DMD.

DETAILED DESCRIPTION:
The study includes a 52-week, randomized, double-blind, placebo-controlled period, followed by a 2-week follow- up. Approximately 125 boys with DMD will be enrolled in this trial, with 2 boys receiving edasalonexent for every 1 boy receiving placebo.

Following completion of the treatment period, patients may elect to continue in a separate open-label extension study.

ELIGIBILITY:
Inclusion Criteria:

* Written consent/assent by patient and/or legal guardian as per regional and/or Institutional Review Board (IRB)/Independent Ethics Committee (IEC) requirements
* Diagnosis of DMD based on a clinical phenotype with increased serum creatine kinase (CK) and documentation of mutation(s) in the dystrophin gene known to be associated with a DMD phenotype
* Able to perform stand from supine without assistance in ≤ 10 seconds
* Able to perform the 10MWT and 4-stair climb
* Followed by a doctor or medical professional who coordinates Duchenne care on a regular basis and willingness to disclose patient's study participation with medical professionals

Exclusion Criteria:

* Use of corticosteroids within 24 weeks prior to Day 1; use of inhaled, intranasal, and topical corticosteroids is permitted
* Use of another investigational drug, idebenone, or dystrophin-focused therapy within 4 weeks. Exception: Patients who have received at least 24 weeks of a stable dose of eteplirsen prior to Day 1, and expected to continue treatment, will be eligible
* Use of the following within 4 weeks prior to Day 1: immunosuppressive therapy, warfarin, phenytoin, S mephenytoin, cyclosporine, dihydroergotamine, ergotamine, fentanyl, alfentanil, pimozide, quinidine, sirolimus, tacrolimus, or paclitaxel
* Use of human growth hormone within 3 months prior to Day 1
* Other prior or ongoing significant medical conditions

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M Donovan, Chief Medical Officer, MD, PhD, Study Chair — Catabasis Pharmaceuticals
Locations (40):
- United States (24):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - UC Davis, Sacramento, California
  - Nemours Children's Hospital, Orlando, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Rush University Children's Hospital, Chicago, Illinois
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - University of Kansas Medical Center, Fairway, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Las Vegas Clinic, Las Vegas, Nevada
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Shriners Hospitals for Children, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Children's Health Queensland Children's Hospital and Health Service, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - London Health Sciences Centre - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- Germany (2):
  - University of Hamburg, Hamburg
  - University of Munich, Munich
- Children's University Hospital, Dublin, Ireland
- Hadassah Medical Center, Jerusalem, Israel
- Queen Silvia Children's Hospital, Gothenburg, Sweden
- United Kingdom (4):
  - Bristol Children's Hospital, Bristol
  - Evelina Children's Hospital, London
  - Great Ormond Street Hospital (GOSH), London
  - Royal Manchester Children's Hospital, Manchester

REFERENCES:
- [Derived] Finkel RS, McDonald CM, Lee Sweeney H, Finanger E, Neil Knierbein E, Wagner KR, Mathews KD, Marks W, Statland J, Nance J, McMillan HJ, McCullagh G, Tian C, Ryan MM, O'Rourke D, Muller-Felber W, Tulinius M, Burnette WB, Nguyen CT, Vijayakumar K, Johannsen J, Phan HC, Eagle M, MacDougall J, Mancini M, Donovan JM; (For the PolarisDMD Study Group). A Randomized, Double-Blind, Placebo-Controlled, Global Phase 3 Study of Edasalonexent in Pediatric Patients with Duchenne Muscular Dystrophy: Results of the PolarisDMD Trial. J Neuromuscul Dis. 2021;8(5):769-784. doi: 10.3233/JND-210689. PMID 34120912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center study conducted by 37 principal investigators at 37 study centers in 8 countries (United States, Canada, United Kingdom, Germany, Ireland, Israel, Sweden, and Australia.)
Pre-assignment Details: A total of 151 patients were screened of which 20 failed screening. 131 patients who participated in the study included 126 randomized patients and 5 participants who were dosed siblings of previously randomized patients.
Period: Overall Study
Arm/Group | Dose 1 | Placebo
Started | 88 | 43
Completed | 85 | 37
Not Completed | 3 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Non-compliance with study drug | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Progressive disease | 1 | 0
Not completed — Withdrawal by parent/guardian | 1 | 0
Not completed — Starting another treatment | 0 | 1
Not completed — noncompliance with study procedures | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All patients who received at least 1 dose of study drug, with patients analyzed based on the actual study treatment received. This included the set of patients who were assigned the same treatment as their randomized sibling.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose 1 | Placebo | Total
Number analyzed (Participants) | 88 | 43 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.65 (1.048) | 5.77 (0.995) | 5.69 (1.029)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 88 | 43 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 6 | 20
  Not Hispanic or Latino | 69 | 35 | 104
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race is missing for one subject.
  A patient who reported more than 1 race was categorized as multiracial.
  Participants
    number analyzed (Participants) | 87 | 43 | 130
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 3 | 2 | 5
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 4 | 1 | 5
    White | 74 | 38 | 112
    More than one race | 3 | 1 | 4
    Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in North Star Ambulatory Assessment (NSAA)
Description: To assess change from baseline in North Star Ambulatory Assessment(NSAA) Total Score at Wk52. NSAA is clinician-reported outcome instrument designed to measure ambulatory function in males with Duchenne muscular dystrophy(DMD). Patients asked to perform 17 different functional activities,including 10MWT,rising from sit to stand,standing on one leg,climbing & descending a step,stand from supine, lifting the head, standing on heels, & jumping. Each function activity will be scored as0=(unable to achieve independently),scored as1=(modified method but achieves goal independent of physical assistance from another),or scored as2=(no obvious modification of activity)or "Not Scored". If NSAA test was performed & any of the individual items are scored as "not scored"(i.e, for reasons unrelated to patients physical capabilities), corresponding total score will be set to missing. Sum of 17 scores will be used to form an ordinal total score(range 0-34).Higher scores imply better functional status
Time Frame: Baseline (Day 1) to Week 52
Population: Full Analysis population: All patients in the Randomized Population who received at least 1 dose of study drug and provided at least 1 valid post Baseline NSAA efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Placebo
Number analyzed (Participants) | 81 | 38
score on a scale | -1.5 (4.41) | -1.8 (3.81)

2. Secondary Outcome: Change From Baseline in 10-meter Walk/Run Test
Description: To assess the changes from baseline to Week 52 on the 10-meter walk/run test (10MWT). For timed function tests (TFTs), the time will be set to 12 seconds and the speed to 0 if the TFT assessment meets the following TFT grading criteria. Grade of 1 or 2 (from a 6-point scale). 1=Unable to walk independently 2=Unable to walk independently but can walk with knee-ankle foot orthoses or support from a person 3=Highly adapted wide based lordotic gait. Cannot increase walking speed 4=Moderately adapted gait. Can pick up speed but cannot run 5=Able to pick up speed, but runs with a double stance phase, i.e. cannot achieve both feet off the ground 6=Runs and gets both feet off the ground (with no double stance phase)
Time Frame: Baseline (Day 1) to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Placebo
Number analyzed (Participants) | 81 | 38
score on a scale | -0.0058 (0.03010) | -0.0093 (0.02538)

3. Secondary Outcome: Change From Baseline in Time to Stand From Supine
Description: To assess the change from baseline in the stand from supine speed at Week 52. For timed function tests (TFTs) , the time will be set to 12 seconds and the speed to 0 if the TFT assessment meets the following TFT grading criteria. Grade of 1 or 2 (from a 6-point scale). 1 = Unable to stand from supine, even with use of a chair, 2 = Assisted Gowers - requires furniture for assist in arising from supine to full upright posture (no time to be recorded) 3=Rolls over, stands up with both hands "climbing up" the legs to achieve full upright posture 4=Rolls over, stands up with 1 hand support on leg 5=Rolls to the side and stands up with one or both hands on the floor to start to rise but does not touch legs 6=Stands up without rolling over or using hands on legs or floor
Time Frame: Baseline (Day 1) to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Placebo
Number analyzed (Participants) | 81 | 38
score on a scale | -0.0389 (0.06728) | -0.0459 (0.06171)

4. Secondary Outcome: Change From Baseline in 4-stair Climb
Description: To assess the change from baseline to Week 52 on the 4-Stair Climb. For timed function tests (TFTs) , the time will be set to 12 seconds and the speed to 0 if the TFT assessment meets the following TFT grading criteria. Grade of 1(from a 6-point scale)1=Unable to climb 4 standard stairs(no time recorded) 2=Climbs 4 standard stairs "marking time"(climbs one foot at a time, with both feet on a step before moving to next step), uses both arms on one or both handrails or uses 1 handrail and the other arm pushes on the leg 3=Climbs 4 standard stairs "marking time", using one arm on one handrail or one hand pushing on leg or body 4=Climbs 4 standard stairs "marking time", not needing handrail and not using hands to push on leg 5=Climbs 4 standard stairs alternating feet, needs handrail/s for support or uses arms to push on the leg or body 6=Climbs 4 standard stairs alternating feet, not needing handrail support or using arm to push on the leg
Time Frame: Baseline (Day 1) to Week 52
Population: Full Analysis Population: All patients in the Randomized Population who received at least 1 dose of study drug and provided at least 1 valid post Baseline NSAA efficacy assessment).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Placebo
Number analyzed (Participants) | 81 | 38
score on a scale | -0.0220 (0.08920) | -0.0392 (0.07352)

5. Secondary Outcome: Safety and Tolerability Measured by Number of Treatment- Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Adverse events that occurred from the time of the administration of the first dose of investigational product (IP) through the end of the safety follow-up were considered treatment-emergent AEs (TEAEs). Serious adverse event (SAE).
Time Frame: Up to Week 52
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Dose 1 | Placebo
Number analyzed (Participants) | 88 | 43
participants
  Treatment Emergent Adverse Event (TEAEs) | 85 | 41
  Related Treatment Emergent Adverse Event (TEAEs) | 61 | 14
  Serious TEAE | 1 | 1
  Serious Related TEAEs | 0 | 0
  TEAEs Leading to Study Discontinuation | 1 | 0
  Treatment-Related TEAEs Leading to Study Discontinuation | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: Subjects with more than one AE of the same system organ class (SOC) / preferred term (PT) were counted only once for that SOC / PT.
Arm/Group | Dose 1 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/88 | 1/43
Other Adverse Events (participants affected / at risk) | 85/88 | 41/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 (N=88) | Placebo (N=43)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose 1 (N=88) | Placebo (N=43)
Diarrhoea (Gastrointestinal disorders) | 54 | 12
Vomiting (Gastrointestinal disorders) | 29 | 11
Abdominal pain upper (Gastrointestinal disorders) | 15 | 9
Nausea (Gastrointestinal disorders) | 7 | 5
Constipation (Gastrointestinal disorders) | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 7 | 1
Abdominal discomfort (Gastrointestinal disorders) | 4 | 1
Dental caries (Gastrointestinal disorders) | 2 | 1
Faeces soft (Gastrointestinal disorders) | 2 | 1
Toothache (Gastrointestinal disorders) | 3 | 0
Nasopharyngitis (Infections and infestations) | 19 | 9
Upper respiratory tract infection (Infections and infestations) | 18 | 5
Ear infection (Infections and infestations) | 7 | 5
Influenza (Infections and infestations) | 10 | 2
Pharyngitis streptococcal (Infections and infestations) | 4 | 4
Gastroenteritis (Infections and infestations) | 3 | 2
Gastroenteritis viral (Infections and infestations) | 3 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 2
Conjunctivitis (Infections and infestations) | 2 | 1
Impetigo (Infections and infestations) | 3 | 0
Tonsillitis (Infections and infestations) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pyrexia (General disorders) | 17 | 9
Fatigue (General disorders) | 6 | 0
Influenza like illness (General disorders) | 0 | 5
Non-cardiac chest pain (General disorders) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 14 | 4
Contusion (Injury, poisoning and procedural complications) | 6 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 20 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 12 | 8
Dizziness (Nervous system disorders) | 3 | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 2 | 1
Weight increased (Investigations) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 6 | 2
Chromaturia (Renal and urinary disorders) | 2 | 2
Pollakiuria (Renal and urinary disorders) | 3 | 0
Ear pain (Ear and labyrinth disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT03703882/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT03703882/SAP_001.pdf